CLINICAL TRIAL: NCT04717089
Title: The Rapid Conversion of Ordinary Recovery Beds to an Overnight Intensive Recovery (OIR) to Alleviate the High Pressure on Postoperative Intensive Care Demands During COVID-19 Pandemics in a Local Tertiary Hospital: a Multi-perspective Value-based Analysis
Brief Title: Extended Post Anaesthetic Care in PACU During COVID-19: Multi-perspective Value-based Analysis
Status: Completed | Type: Observational
Sponsor: Tuen Mun Hospital (Other Government)
Collaborators: Anaesthesia & Operation Theatre Service, Tuen Mun Hospital, Hong Kong (Unknown); Intensive Care Unit, Tuen Mun Hospital, Hong Kong (Unknown)
Responsible Party: Principal Investigator, Lau Hon Wai, Medical Officer, Tuen Mun Hospital
Other Study IDs: TMH-ExRR-001
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Overnight Intensive Recovery; Postoperative Care
MeSH Terms: interventions — Recovery Room

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postoperative patients admitted to TMH extended post anaesthetic care in PACU: Exclusion criteria:
  * Patients awaiting ICU admission in the ordinary recovery room
  * Patients requiring level 3 intensive care on arrival at the recovery room
  Interventions: Other: overnight intensive recovery / extended post anaesthetic care in PACU
- Postoperative patient admitted to ICU with case matched: Inclusion criteria:
  o Based on case matched with the extended post anaesthetic care in PACU

INTERVENTIONS:
Other: overnight intensive recovery / extended post anaesthetic care in PACU — From January 2020, during COVID-19 first pandemics in Hong Kong, a bundle of interim measures was implemented with the joint efforts of the Department of Anaesthesia and Operating Theatre Services (A&OT) and Intensive Care Unit (ICU), and two ordinary recovery beds were converted into extended post anesthetic care in PACU (ExRR), based on the concept of overnight intensive recovery (OIR) to provide level 2 intensive care to patients undergoing major or ultra-major operations or having multiple comorbidities warranted intensive care in the immediately postoperative periods. This was conducted over 3 pandemic waves in Hong Kong.
  Groups: postoperative patients admitted to TMH extended post anaesthetic care in PACU

SUMMARY:
To evaluate the value-based effectiveness of the implementation of TMH Extended post anaesthetic care in PACU during COVID-19 pandemics by an institutional matched case-control and quantitative survey study Two ordinary recovery beds were converted to an overnight intensive recovery ("Extended post-anesthetic care in PACU") within the operating theatre complex of Tuen Mun Hospital during COVID-19 pandemics, in an attempt to free the ICU bed and resources from postoperative patients. This study was designed to evaluate the efficacy and staff perceptions towards the abrupt implementation of TMH extended post-anesthetic care in PACU by mobilization of the existing OT resources to cope with the COVID-19 emergency situations. The value-based analysis would look into the implementation effectiveness in twofold: 1) the clinical efficacy using a case-control audit on clinical outcomes and 2) the staff acceptance by means of the staff attitudes survey. Hopefully, this would provide a multi-perspective evaluation of the implementation strategies and aid planning of new services in the future.

DETAILED DESCRIPTION:
2 parts are included in this study

The Matched Case-Control study, with the aim of analyzing the clinical efficacy of TMH Extended post-anesthetic care in PACU during COVID-19 in a value-based healthcare model. We included all postoperative patients admitted in TMH Extended post-anesthetic care in PACU during COVID epidemics, excluding patients awaiting ICU in the ordinary recovery room or patients requiring level 3 intensive care on arrival in the recovery room. Three activation periods of 水xtended post-anesthetic care in PACU service (10 Feb - 26 Apr 2020 / 27 Jul - 13 Sep 2020 / 14 Dec 2020 - 28 Feb 2021), and performed case matching with the postoperative patient with similar clinical characteristics entering intensive care unit directly in recent 10 years, with each case matched with specifically 5 control. We evaluate the value-based health care efficacy, including the amount of healthcare expenditure based on bed occupancy and manpower, rate of elective discharge to intensive care unit from extended post-anesthetic care in PACU, rate of unanticipated intensive care admission within 48hrs upon discharge to the general ward, and length of hospital stay, and the total number of ICU bed spared.

The staff attitude survey, with the aim to investigate the staff perception towards the implementation of TMH extended post-anesthetic care in PACU during COVID-19 pandemics based on the Technology Acceptance Model in healthcare. We designed a questionnaire based on Technology Acceptance Model, and distributed it to medical and nursing staff involved in extended post anaesthetic care in PACU service, and evaluate the perceived usefulness, perceived ease of use, social influence of subjective norm, and perceived behavioral control of facilitating condition. A differential analysis would be conducted for the evaluation.

ELIGIBILITY:
Inclusion criterion:

o Postoperative patients admitted to TMH Extended post anesthetic care in PACU during COVID-19 pandemics

Exclusion criteria:

* Patients awaiting ICU admission in the ordinary recovery room
* Patients requiring level 3 intensive care on arrival at the recovery room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: o The operation periods of TMH Extended post anesthetic care in PACU during COVID-19 and therefore the number of cases included in this study was largely bound by the administrative decision of hospital management based on the ICU bed pressure during COVID-19 situations. All patients being admitted to TMH Extended post anesthetic care in PACU during the three periods of service activation amid COVID-19 pandemics, i.e. from 10 February 2020 to 26 April 2020, from 27 July 2020 to 13 September 2020, from 14 December 2020 to 28 February 2021 were included in this audit. To increase the statistical power above 0.8, a control-to-case ratio of 5 will be adopted for case matching based on the assumption of having the correlation coefficient greater than 0.2 or the prevalence of exposure in the control group less than 0.15.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
total number of ICU bed days spared | during study period, up to 1 year

SECONDARY OUTCOMES:
amount of healthcare expenditures based on bed occupancy and manpower | during study period, up to 1 year
number of unanticipated intensive care unit admission within 48 hours upon discharge to general ward | 48 hour
rate of elective discharge to the intensive care unit | After extended post anaesthetic care in PACU service by case. Up to 24 hour
length of hospital stays | during admission or patient death, typically up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Lam, Study Director — Tuen Mun Hospital
Locations (1):
- Tuen Mun Hospital, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No